CLINICAL TRIAL: NCT00580138
Title: Real-Time Internet Evaluation of Oropharyngeal Dysphagia
Brief Title: Real-Time Internet Evaluation of Swallowing
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Collaborators: University of Illinois at Chicago (Other); University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 1R01DC005603 (NIH); 1R01DC005603 (NIH)
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Results first posted 2010-06-07 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-01

CONDITIONS: Head and Neck Cancer; Stroke
Keywords: Deglutition Disorders; Evaluation; Real-time internet
MeSH Terms: conditions — Head and Neck Neoplasms; Stroke; Deglutition Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stroke or Head & Neck Cancer: Any subject who has suffered a stroke or has some form of head & neck cancer (non-laryngectomee) may be enrolled.

SUMMARY:
The purpose of this study is to determine whether real-time internet evaluations of swallowing, or x-ray swallow studies viewed over closed internet circuit, are a reliable method of evaluating swallowing function.

DETAILED DESCRIPTION:
The objective of this proposal is to establish the validity of an Internet based protocol for real-time, remote, telefluoroscopic evaluation of oropharyngeal swallowing function. The investigators will achieve this goal by testing the hypothesis that oropharyngeal swallowing function evaluated by an experienced speech-language pathologist (SLP) using a remote, interactive, real-time, dynamic Internet telefluoroscopic procedure, which was developed in the PI's laboratory, has an acceptable level of agreement with the evaluations performed by an experienced SLP who is present in the fluoroscopy suite and using the traditional videofluoroscopic methodology. In other words, the primary aim of this investigation is to determine whether the telemedicine approach to evaluation of swallowing function is reliable relative to the traditional method by which a clinician is in direct contact with a patient for a pre-examination interview, clinical examination, and videofluoroscopic evaluation of swallowing function. Confirmation of the reliability of the telefluoroscopic evaluation of oropharyngeal dysphagia (hereafter referred to as dysphagia) can result in equity of access for underserved groups for whom SLPs with expertise in evaluating swallowing function are locally unavailable. Ultimately, the success of this project could translate specialty services into routine clinical practice across the United States and globally.

ELIGIBILITY:
Inclusion Criteria:

* Stroke, Head & neck cancer, referred for swallowing evaluation.

Exclusion Criteria:

* No stroke or no head and neck cancer, or not referred for swallowing evaluation.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who have suffered a stroke and/or head and neck cancer and are referred for evaluation of swallowing function.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2005-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne Perlman, Principal Investigator — University of Illinois, Urbana Champaign; Gary H McCullough, Ph.D., Principal Investigator — UAMS Medical Center
Locations (2):
- United States (2):
  - University of Illinois, Urbana-Champaign, Illinois
  - University of Wisconsin, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stroke or Head & Neck Cancer
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Stroke or Head & Neck Cancer
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (4)
Gender [Count of Participants; unit: Participants]
  Female | 13
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Reliability Ratings Among Clinicians Using Real-time Internet Evaluation of Swallowing.
Description: Percentages were calculated for agreement between ratings made by on site clinician and clinician off site with telemedicine.
Time Frame: 2 years
Measure: Number; unit: percent agreement
Arm/Group | Stroke or Head & Neck Cancer
Number analyzed (Participants) | 30
percent agreement | 60

ADVERSE EVENTS:
Arm/Group | Stroke or Head & Neck Cancer
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No